CLINICAL TRIAL: NCT00107848
Title: A 1 Year Open Label, Flexible Dosage Extension Study to Assess the Safety and Continued Effectiveness of PROVIGIL® (Modafinil) Treatment in Children and Adolescents With Excessive Sleepiness Associated With Narcolepsy or Obstructive Sleep Apnea/Hypopnea Syndrome
Brief Title: PROVIGIL® (Modafinil) Treatment in Children and Adolescents With Excessive Sleepiness Associated With Narcolepsy or Obstructive Sleep Apnea/Hypopnea Syndrome
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Cephalon (Industry)
Organization: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Allocation: Non-Randomized | Model: Single Group | Purpose: Treatment
Other Study IDs: C1538/3029/ES/MN-Open label
Record Dates: First submitted 2005-04-08; First posted 2005-04-11 (Estimated); Last update posted 2014-05-09 (Estimated); Status verified 2014-05

CONDITIONS: Narcolepsy; Sleep Apnea, Obstructive
Keywords: Pediatric Narcolepsy; Pediatric OSA; CPAP; Pediatric Narcolepsy or OSAHS
MeSH Terms: conditions — Narcolepsy; Sleep Apnea, Obstructive | interventions — Modafinil

INTERVENTIONS:
Drug: Modafinil

SUMMARY:
The primary objective of the study is to evaluate the safety and tolerability of treatment with PROVIGIL in children and adolescents with excessive sleepiness (ES) associated with narcolepsy or OSAHS (obstructive sleep apnea/hypopnea), when administered for up to 12 months. Safety and tolerability will be evaluated throughout the study by means of adverse event information, clinical laboratory test results, vital signs measurements, and body weight and height measurements; quarterly physical examination findings; and 12 lead electrocardiograph (ECG) evaluations at the end of the study. In addition, the cognitive and behavioral effects of PROVIGIL will be assessed quarterly as measured by the Child Behavior Checklist for Ages 6-18 (CBCL/6-18), a brief psychiatric interview, and the Kaufman Brief Intelligence Test (KBIT 2).

DETAILED DESCRIPTION:
PROVIGIL is a registered trademark of Genelco, S.A., licensed to Cephalon, Inc.

ELIGIBILITY:
Inclusion Criteria:

* Appropriate written assent is obtained from the patient and written informed consent is obtained from the parent or legal guardian (defined by the IEC/IRB)
* A boy or girl aged 6 through 16 years (at the start of the previous double blind study), inclusive, who participated in study C1538/3027/NA/MN or C1538/3028/AP/MN
* Have a diagnosis (as established in the previous double blind study) of narcolepsy (or presumed narcolepsy) or OSAHS according to the criteria established by the International Classification of Sleep Disorders (ICSD) manual of the American Academy of Sleep Medicine (AASM)
* Continue to be in good health as determined by a medical and psychiatric history, ECGs, physical examination findings, serum chemistry, hematology, and urinalysis
* Have blood pressure values greater than those for the 5th percentile and less than the 95th percentile on the National High Blood Pressure Education Program guidelines for blood pressure levels for boys and girls ages 6 through 16 years
* Girls who are post menarche or sexually active who have a negative urine pregnancy test at the screening/baseline visit, must be using a medically acceptable method of birth control, and must agree to continued use of this method for the duration of the study (and for 30 days after participation in the study). Acceptable methods of birth control include: barrier method with spermicide; steroidal contraceptives (oral, topical [patch], implanted, and injected) in conjunction with a barrier method; intrauterine device (IUD); or abstinence
* No positive urine drug screen (UDS) for any illicit drug or alcohol (ethanol) at baseline visit, unless a false positive is suspected, in which case the UDS will be repeated. If the patient has a positive drug screen for methylphenidate or amphetamine at screening, the patient must have a negative UDS after a washout period and prior to baseline.
* Have a parent or legal guardian who is willing to participate in the study
* Continue to meet inclusion criteria from the previous study, as appropriate

Exclusion Criteria:

* Have self induced sleep deprivation/poor sleep hygiene
* Have a past or present seizure disorder (except history of a single febrile seizure), a history of psychosis, or of clinically significant head trauma (eg, brain damage) or past neurosurgery
* Have a history of suicide attempt, or are at suicidal risk
* A clinically significant drug sensitivity to stimulants such as amphetamine, dextroamphetamine, methylphenidate, or pemoline; and modafinil or any of its components
* Any disorder that could interfere with drug absorption, distribution, metabolism, or excretion (including previous gastrointestinal surgery)
* Active, clinically significant gastrointestinal, cardiovascular, hepatic, renal, hematologic, neoplastic, endocrine, neurologic, immunodeficiency, pulmonary, or other major clinically significant disorder/disease
* Any clinically significant deviation from the normal range(s) in the ECG or physical examination findings, or clinical laboratory (ie, hematology, serum chemistry, urinalysis) test results at the screening/baseline visit
* Absolute neutrophil count (ANC) below the lower limit of normal at the baseline visit (NOTE: If the ANC is below the lower limit of normal at the baseline visit, the medical monitor will be consulted for continued eligibility in the study.)
* A seated pulse outside the range of 60 through 115 bpm after resting for 5 minutes
* A total daily intake of more than 500 mg of caffeine per day (eg, approximately ten 12 ounce caffeinated sodas, 5 cups of coffee or tea, or about 25 ounces of chocolate per day) within 1 week of the baseline visit
* Pregnant or lactating/nursing; any child who becomes pregnant during the study will be withdrawn.

Ages: 6 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 280
Dates: Start 2004-10; Study Completion 2005-09

PRIMARY OUTCOMES:
The primary objective of the study is to evaluate the safety and tolerability of treatment with PROVIGIL in children and adolescents with excessive sleepiness (ES) associated with narcolepsy or OSAHS, when administered for up to 12 months.

SECONDARY OUTCOMES:
The secondary objective of the study is to evaluate long-term effectiveness by using: the Clinical Global Impression of Change (CGI C) ratings for severity of ES and the total score from the Pediatric Daytime Sleepiness Scale (PDSS)

CONTACTS AND LOCATIONS:
Locations (61):
- United States (55):
  - Robert Doekel, Jr., M.D., Birmingham, Alabama
  - Chris M. Makris, M.D., Birmingham, Alabama
  - Barbara Harris, Ph.D., Phoenix, Arizona
  - Derek Loewy, Ph.D., Tucson, Arizona
  - Joseph McCarty, M.D., Fort Smith, Arkansas
  - Samuel Boellner, M.D., Little Rock, Arkansas
  - Julie Thompson-Dobkin, D.O., Huntington Beach, California
  - Mark Buchfuhrer, M.D., Long Beach, California
  - Yury Furman, M.D., Los Angeles, California
  - Stuart Menn, M.D., Palm Springs, California
  - Lawrence Sher, M.D., Rolling Hills Estates, California
  - Milton K. Erman, M.D., San Diego, California
  - Jed Black, M.D., Stanford, California
  - Edward O'Malley, Norwalk, Connecticut
  - Elias H. Sarkis, Gainesville, Florida
  - Americo Padilla, M.D., Miami, Florida
  - Martin A. Cohn, M.D., Naples, Florida
  - D. Alan Lankford, Ph.D., Atlanta, Georgia
  - Gary Montgomery, M.D., Atlanta, Georgia
  - Jerry Silverboard, M.D., Atlanta, Georgia
  - Charles Wells, Jr., M.D., Macon, Georgia
  - Joel Greenberg, Savannah, Georgia
  - Robert M. Cohen, Stockbridge, Georgia
  - Stephen H. Sheldon, D.O., FAAP, Chicago, Illinois
  - Michael Kohrman, M.D., Chicago, Illinois
  - James Cook, M.D., Danville, Indiana
  - William Leeds, D.O., Topeka, Kansas
  - Karen Waters, M.D., Louisville, Kentucky
  - Margaret Ann Springer, M.D., Shreveport, Louisiana
  - Helene A. Emsellem, M.D., Chevy Chase, Maryland
  - Marc Raphaelson, Frederick, Maryland
  - George Zureikat, M.D., Flint, Michigan
  - John Harsh, Ph.D., DABSM, Hattiesburg, Mississippi
  - William Torch, M.D., MS, Reno, Nevada
  - Kathleen Ryan, M.D., Mount Laurel, New Jersey
  - Monroe Karetzky, M.D., Newark, New Jersey
  - Lee Brooks, M.D., Princeton, New Jersey
  - Marc Seelagy, M.D., Trenton, New Jersey
  - Gary Zammit, M.D., New York, New York
  - Carol Rosen, Cleveland, Ohio
  - Michael Neeb, Ph.D., Toledo, Ohio
  - Ramalinga Reddy, Toledo, Ohio
  - William C. Orr, Ph.D., Oklahoma City, Oklahoma
  - Jorg Pahl, M.D., Oklahoma City, Oklahoma
  - Judith Owens, M.D., MPH, Providence, Rhode Island
  - Richard Bogan, M.D., FCCP, Columbia, South Carolina
  - Julie Jacques, D.O., Morristown, Tennessee
  - John Hudson, M.D., Austin, Texas
  - David Sperry, M.D., Dallas, Texas
  - Todd J. Swick, M.D., Houston, Texas
  - Jerry J. Tomasovic, M.D., San Antonio, Texas
  - Radiant Research, Salt Lake City, Salt Lake City, Utah
  - James M. Ferguson, M.D., Salt Lake City, Utah
  - James Perlstrom, Fairfax, Virginia
  - Robert J. Reichler, Seattle, Washington
- Canada (6):
  - Adam Moscovitch, M.D., Calgary, Alberta
  - Manisha Witmans, Edmonton, Alberta
  - Lawrence Reinish, Parry Sound, Ontario
  - Leonid Kayumov, M.D., Scarborough Village, Ontario
  - Mortimer Mamelak, M.D., Toronto, Ontario
  - Colin Shapiro, Ph.D., Toronto, Ontario